CLINICAL TRIAL: NCT00317720
Title: Phase I-II Study of Trastuzumab in Combination With RAD001 in Patients With HER-2 Overexpressing, PTEN-deficient Metastatic Breast Cancer Progressing on Trastuzumab-Based Therapy
Brief Title: Trastuzumab and RAD001 in Patients With Human Epidermal Growth Receptor 2 (HER-2) Overexpressing Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0471
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: Breast Cancer; Metastatic Breast Cancer; Trastuzumab; RAD001; Herceptin
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Trastuzumab; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Trastuzumab + RAD001 (Experimental): Trastuzumab loading dose is 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle. Starting RAD001 dose 10 mg by mouth daily.
  Interventions: Drug: Trastuzumab; Drug: RAD001

INTERVENTIONS:
Drug: Trastuzumab — Loading dose = 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle.
  If participant on trastuzumab at time of registration, loading dose deferred and received maintenance dose (6 mg/kg every 3 weeks). If the last trastuzumab dose was given 1 week (for participants receiving 2 mg/kg/week), or 3 weeks before registration (for participants receiving 6 mg/kg every 3 weeks), a loading dose (8 mg/kg) was given followed by maintenance dose.
  Other Names: Herceptin
Drug: RAD001 — Starting dose 10 mg by mouth daily. Phase I dose finding from two dose levels of daily RAD001 (5 and 10 mg).
  Other Names: Everolimus

SUMMARY:
Primary Objectives:

1. To identify the optimal dose and pharmacokinetics of RAD001 in combination with trastuzumab in a Phase I trial
2. To determine the efficacy of RAD001 plus trastuzumab in HER-2-overexpressing patients with resistance to trastuzumab-based therapy for metastatic breast cancer in a Phase II trial.

   1. Trastuzumab resistance will be defined as the development of progressive disease after trastuzumab-based therapy for metastatic breast cancer. Patients who develop metastases while receiving adjuvant or neoadjuvant trastuzumab will be eligible.
   2. Efficacy would be measured by the rate of objective response plus stable disease lasting 6 months (complete response (CR) + partial response (PR) + stable disease SD).

Secondary objectives:

1. To determine the pharmacokinetics of RAD001 in combination with trastuzumab. In the phase II portion of the study, pharmacokinetic studies will be optional.
2. To determine the nature and degree of toxicity of RAD001 in combination with trastuzumab in this cohort of patients
3. To determine expression levels of total and phosphorylated mTOR and p70S6K-T389-P as well as relevant downstream signaling components (e.g., S6, 4E-BP1) in pre- and post- treatment tumor samples.
4. To correlate biomarker expression with response to therapy.

DETAILED DESCRIPTION:
RAD001 is a new drug that was designed to block proteins that are important in the development and growth of cancer. It may also stop the growth of new blood vessels that help tumor growth, resulting in cell death.

Trastuzumab is a monoclonal antibody that binds to the HER-2 molecule on the surface of cancer cells. It does not bind to cells that do not have the HER-2 molecule. Trastuzumab slows the growth of cancer cells and also makes them more able to be treated with other chemotherapy drugs.

Before you begin to receive the study drug, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study. You will have your complete medical history recorded, and a physical exam, including measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate) will be performed. Routine blood tests (about 2 teaspoons) will be collected within 1 week before therapy. Cancer tissue taken at the time of your initial diagnosis or surgery will be collected. Special stains will be done that will help find ways in which researchers can predict the response of your cancer to trastuzumab plus RAD001. Women who are able to have children must have a negative urine pregnancy test. Some participants may need x-rays and/or positron emission tomography (PET) scans before receiving study drug and again within 3 weeks after the start of therapy.

If you are found to be eligible to take part in this study, you will receive RAD001 tablets by mouth once a day. Every 3 weeks (21 days) is considered 1 course of the study. The dose of trastuzumab you receive on this study will not be different from what you were receiving before this study started.

If you are participating in the Phase I portion of the study, you will have about 4 teaspoons of blood drawn before you start the study on Day 1. Blood samples will be drawn prior to initiation of treatment and at 0.5, 1, 2, 5, 8, 24 hours. You will also have around 4 teaspoons of blood drawn on Day 15 (before the start of treatment and at 0.5, 1, 2, 5, 8, and 24 hours).

While on study, you will have weekly blood tests (about 2 teaspoons) for the first 3 weeks. After 3 weeks, if you tolerate the study drug well, your blood tests (about 2 teaspoons each time) will be drawn once every 3 weeks, or as often as your physicians feel that they are necessary. Six (6) weeks after your first cycle of study drug, you will undergo x-rays, computed tomography (CT) scans, magnetic resonance imaging (MRI), or PET scans to see how you are responding to the study drug. If the disease shows a response to the study drug or is stable, then future x-rays, CT scans, MRI or PET scans will be performed every 6 weeks, or as often as the physician feels it is necessary. After that, the scans will be performed every 9 weeks, or as often as the physician feels it is necessary. A physical exam, including vital signs (blood pressure, heart rate, temperature, and breathing rate), will be done every 3 weeks and any time the physician feels it is necessary.

You will continue to take the study drug as long as you continue to benefit from it. You may be removed from this study if you do not respond after 2 courses of the study drug, intolerable side effects occur, or the disease gets worse. Your dose may be lowered if certain side effects occur.

Once you come off study, a physical exam, measurement of vital signs (blood pressure, heart rate, temperature, and breathing rate), a blood test (about 2 teaspoons), x-rays, and/or scans will be done.

This is an investigational study. Trastuzumab is commercially available for use as a single therapy or in combination with paclitaxel. However, the combination of trastuzumab and RAD001 is experimental. The FDA has authorized RAD001 for use in research only. Up to 47 patients will take part in this multicenter study. Up to 36 will be enrolled at UT MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. History of biopsy-proven HER-2-overexpressing breast cancer and radiographic evidence of metastatic disease. The HER-2 status can be determined either by immunohistochemistry (score, 3+) or by fluorescence in situ hybridization.
2. History of trastuzumab resistance, defined as the development of progressive disease after trastuzumab-based therapy for metastatic breast cancer. Patient may not have received more than 2 prior trastuzumab-based regimens and one lapatinib-based regimen (either as single agent or in combination with chemotherapy)for metastatic breast cancer. Patients who develop metastatic disease during or after adjuvant or neoadjuvant trastuzumab are eligible.
3. Performance status 0-2 (by Eastern Cooperative Oncology Group (ECOG) scale).
4. Absolute neutrophil count (ANC) 1500/µl or higher; Platelets 100,000/µl or higher; Hemoglobin 9.0 gm/dL or higher; Serum creatinine 2.0 mg/dL or lower; Total bilirubin 1.5 mg/dL or lower; Serum glutamic pyruvic transaminase (SGPT) up to 3* upper limit of normal; Alkaline phosphatase up to 3* upper limit of normal; Calcium 11.0 mg/dL or lower.
5. Age 18 years or older.
6. Patients must not be pregnant. A pregnancy test will be obtained if the patient is a woman of child-bearing potential, defined as a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months (i.e., who has had menses at any time in the preceding 24 consecutive months).
7. Patients must have signed an informed consent document stating that they understand the investigational nature of the proposed treatment.
8. Patients must have measurable disease using Response Evaluation Criteria in Solid Tumors (RECIST). Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension with longest diameter >/= 20 mm using conventional techniques or >/= 10 mm with spiral computed tomography (CT) scan.
9. Patients may not be receiving any other investigational agents, and must not have received investigational agents within 15 days of enrollment.
10. Left ventricular ejection fraction determined by echocardiogram or multigated acquisition (MUGA) (cardiac scan) must be 50% or higher.

Exclusion Criteria:

1. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
2. Prior treatment with any investigational drug within the preceding 15 days
3. Chronic treatment with systemic steroids or another immunosuppressive agent
4. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases, and patients diagnosed with brain mets or leptomeningeal disease (LMD) within 3 months.
5. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
6. A known history of HIV seropositivity
7. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of RAD001 (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
8. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication (except low dose coumadin)
9. Patients who have received prior treatment with an mTor inhibitor.
10. History of noncompliance to medical regimens.
11. Patients unwilling to or unable to comply with the protocol.
12. Patients who are receiving any other investigational agents
13. Patients exhibiting confusion, disorientation, or having a history of major psychiatric illness that may impair the understanding of the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Esteva, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Result] Morrow PK, Wulf GM, Ensor J, Booser DJ, Moore JA, Flores PR, Xiong Y, Zhang S, Krop IE, Winer EP, Kindelberger DW, Coviello J, Sahin AA, Nunez R, Hortobagyi GN, Yu D, Esteva FJ. Phase I/II study of trastuzumab in combination with everolimus (RAD001) in patients with HER2-overexpressing metastatic breast cancer who progressed on trastuzumab-based therapy. J Clin Oncol. 2011 Aug 10;29(23):3126-32. doi: 10.1200/JCO.2010.32.2321. Epub 2011 Jul 5. PMID 21730275
- See also: The University of Texas (UT) MD Anderson Cancer Center official website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a a pooled analysis, stemming from two Phase I/II trials that occurred concurrently under separate investigational new drug applications (INDs) at The University of Texas MD Anderson Cancer Center (MDACC; IND 69277); and Beth Israel Deaconess Medical Center (BIDMC, IND 76179) with Dana-Farber Cancer Institute (DFCI), May 2006 to May 2009.
Pre-assignment Details: Results data for the two aforementioned BIDMC/DFCI and MDACC trials were combined in order to statistically complete the clinical trials. There were forty participants registered at MDACC, and eleven participants registered at BIDMC/DFCI. Of the eleven participants recruited at BIDMC/DFCI, four were ineligible.
Groups:
- MDACC Trastuzumab + RAD001: Phase I: Trastuzumab loading dose is 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle. RAD001 (Everolimus) 10 mg orally (PO) daily.
  Phase II: RAD001 10 mg/kg daily + Trastuzumab 6 mg/kg maintenance dose
  ClinicalTrials.gov ID: NCT00317720
- BIDMC/DFCI Trastuzumab + RAD001: Phase I: Trastuzumab loading dose is 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle. RAD001 5 or 10 mg by mouth daily.
  Phase II: RAD001 10 mg/kg daily
  ClinicalTrials.gov ID NCT00458237
Period: Overall Study
Arm/Group | MDACC Trastuzumab + RAD001 | BIDMC/DFCI Trastuzumab + RAD001
Started | 40 | 7
Completed | 40 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants were pooled from 2 separate clinical trials (MDACC ClinicalTrials.gov ID NCT00317720) and (BIDMC/DFCI ClinicalTrials.gov ID NCT00458237)
Groups:
- Trastuzumab + RAD001: Trastuzumab loading dose is 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle. RAD001 10 mg given orally daily.
Arm/Group | Trastuzumab + RAD001
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 50 [28 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Hormone receptor status [Number; unit: Participants] — Pathological determination of hormone receptor status, Hormone receptor-positive (estrogen receptor-positive (ER+)/progesterone receptor-positive (PR+)) breast cancers have many hormone receptors. Hormone receptor-negative (estrogen receptor-negative (ER-)/progesterone receptor-negative (PR-)) breast cancers have few or no hormone receptors.
  Participants
    ER or PR positive | 28
    ER and PR Negative | 19
Prior lines of trastuzumab-containing chemotherapy for metastatic breast cancer (MBC) [Number; unit: Participants] — Number of trastuzumab-containing chemotherapy regimens participants had for MBC before starting study
  Participants
    0 | 10
    1 | 29
    2 | 8

OUTCOME MEASURES:

1. Primary Outcome: Optimal Dose of RAD001 in Combination With Trastuzumab (Phase I)
Description: In Phase I, two dose levels of RAD001 were studied: 10 mg (dose level 1) and 5 mg (dose level -1) where each dose was evaluated after cycle 1. At MDACC, the Continual Reassessment Method (CRM) for determining Maximum Tolerated Dose (MTD) was applied to the two predefined RAD001 dose levels; and at DFCI/BIDMC, a 3 x 3 study design was utilized.
  Optimal dose defined as the dose most closely associated with a toxicity rate of 0.20, and toxicity defined as any grade 3 or 4 toxicity (based on Common Terminology Criteria (CTC) version 3.0 except fatigue. Participants underwent clinical evaluation every 3 weeks (one cycle) and radiologic evaluations every 6 weeks. After the second cycle, participants underwent a radiologic evaluation using the same imaging technique used at initial evaluation (ie, computed tomography or magnetic resonance imaging).
Time Frame: Following two 3 week cycles of therapy
Population: At MDACC, sixteen participants total treated at 10 mg (dose level 1) in the Phase I portion of the study with the remainder thirty-four registered in Phase II. At DFCI/BIDMC, the first three participants were included in the Phase I portion of the study, the remaining four of seven registered were in Phase II.
Measure: Number; unit: mg
Groups:
- Trastuzumab + RAD001: Trastuzumab loading dose is 8 mg/kg daily; maintenance dose = 6 mg/kg once per 21 day cycle. RAD001 10 mg PO (by mouth) daily.
Arm/Group | Trastuzumab + RAD001
Number analyzed (Participants) | 19
mg | 10

2. Primary Outcome: Clinical Benefit Response Rate (CBR)
Description: Efficacy measured by the clinical benefit response rate (CBR), defined as confirmed Complete Response (CR) plus Partial Response (PR) at any time plus Persistent Stable Disease (pSD). Confirmed CR is defined as disappearance of all target lesions at the time of radiographic evaluation; pSD was defined as SD lasting 24 weeks. Complete Response (CR): disappearance of all target lesions, and Partial Response (PR): at least a 30% decrease in the sum of longest diameter (LD) of target lesions taking as a reference the baseline sum LD. Stable Disease (SD): neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease taking as references the smallest sum LD since the treatment started.
Time Frame: 6 weeks
Measure: Number; unit: percentage of partcipants
Arm/Group | Trastuzumab + RAD001
Number analyzed (Participants) | 47
percentage of partcipants
  CBR | 34
  CR | 0
  PR | 15
  pSD | 19

ADVERSE EVENTS:
Time Frame: Adverse events assessments graded according to National Cancer Institute Common Toxicity Criteria for Adverse Events, version 3.0 were performed at 3-week intervals and treatment completion. Overall study period was 3 years and 4 months.
Description: Analysis including Adverse Event reporting was pooled for the two Phase I/II trials: MDACC ClinicalTrials.gov ID: NCT00317720; and BIDMC with DFCI ClinicalTrials.gov ID NCT00458237.
Arm/Group | Trastuzumab + RAD001
Serious Adverse Events (participants affected / at risk) | 47/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab + RAD001 (N=47)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 9 (9)
Fatigue (General disorders) | 9 (9)
Hyperglycemia (General disorders) | 13 (13)
Hypokalemia (General disorders) | 6 (6)
Hyperlipidemia (General disorders) | 4 (4)
Infection (General disorders) | 4 (4)
Mucositis (General disorders) | 9 (9)
Transaminitis (General disorders) | 2 (2)
Thrombosis/embolism (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab + RAD001 (N=47)
Anemia (Blood and lymphatic system disorders) | 17 (17)
Lymphopenia (Blood and lymphatic system disorders) | 13 (13)
Neutropenia (Blood and lymphatic system disorders) | 13 (13)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (6)
Fatigue (General disorders) | 23 (23)
Hyperglycemia (General disorders) | 9 (9)
Hypokalemia (General disorders) | 6 (6)
Hyperlipidemia (General disorders) | 9 (9)
Infection (General disorders) | 19 (19)
Mucositis (General disorders) | 25 (25)
Rash (Skin and subcutaneous tissue disorders) | 9 (9)
Transaminitis (General disorders) | 9 (9)

LIMITATIONS AND CAVEATS:
Trial Results were combined for the 2 trials at MDACC & BIDMC/DFCI with US Food & Drug Administration approval for completion with adequate power. As results were pooled for analytic purposes, BIDMC/DFCI protocol was amended to match MDACC protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No